CLINICAL TRIAL: NCT01836965
Title: Replication of the The Multi-Media Social Skills Project for Adolescents With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Michael Murray, MD, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42565EP
Record Dates: First submitted 2013-03-28; First posted 2013-04-22 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Autism Spectrum Disorders
Keywords: Aspergers; Social Skills; Adolescents; High-functioning Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Social Skills Intervention (Experimental): The intervention is a 12-week social skills training program that will consist of a 90 minute group therapy session followed by a 90 minute peer generalization session (in the form of a photography class with typically developing peers) meeting once per week. Each cohort will consist of 6 adolescents with Aspergers or high-functioning autism, who will be joined by 6 typically-developing peers for the photography class. During the group therapy session adolescents will discuss and watch video clips addressing social skills topics relevant to their age group. They will have a chance to practice these skills when paired with a typically developing peer for the photography class.
  Interventions: Behavioral: Social Skills Intervention

INTERVENTIONS:
Behavioral: Social Skills Intervention — Twelve week manual based social skills curriculum targeting social fluency and responsiveness.

SUMMARY:
The objective of this study is to validate a social skills training program manual for adolescents (ages 13-17) with Asperger's Syndrome or high functioning autism. Approximately 150 adolescents with autism spectrum disorders will participate in this study, in groups consisting of 6 adolescents and 6 peer volunteers. Participants will participate in both group therapy and peer generalization sessions (in the form of a photography class) once a week over the course of twelve weeks. Participants and their parents will complete paper and pencil, online, or phone measures and video-recordings to assess the participant's social skills prior to the intervention, at completion of the intervention and three months later.

DETAILED DESCRIPTION:
This study is a pre-test, post-test single group design with post test measures at one week after completion of intervention and follow-up at three months. Approximately 300 adolescents will participate in this study. The study will be conducted in ten cohorts of 12. Each cohort will have 6 participants and 6 adolescent volunteers (peers). Cohorts will be run in a time sequential manner with up to four cohorts running at a time. Participants and their parents will complete pre-test measures including both paper and pencil, online, or phone measures and a video-recording to assess the participant's social interaction skills and fluency. These adolescents will participate in both group therapy and peer generalization sessions once a week over the course of twelve weeks. Upon completion of the intervention, participants and parents will complete paper and pencil, online, or phone measures and video post-test measures. Participants will be encouraged to participate in a follow-up session where the paper and pencil and video measures will be completed again.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 17 years of age
* Must be a Pennsylvania resident
* A primary diagnosis of Asperger's Syndrome or high-functioning autism, as confirmed by the Checklist for Autism Spectrum Disorders (CASD; Mayes, 2012)
* English as primary language spoken
* Ability to fluently speak in full sentences
* A verbal IQ of 85 or above on the Kaufman Brief Intelligence Test, Second Edition(KBIT-2; Kaufman & Kaufman, 1990)

Exclusion Criteria:

* A significant language delay
* Difficulty with aggression directed at peers
* A primary thought disorder
* A secondary disorder of anxiety or depression so severe as to prevent the individual's participation in the treatment
* Low social motivation demonstrated through formalized assessment and/or by responses given to screening interviews assessing treatment goals

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Social Responsiveness Scale Score after Intervention | One Week Post-Intervention
  The Social Responsiveness Scale is a 65 - item survey designed to measure social competence.
Video recording of Social Interaction | One Week Post-Intervention
  Participants will be filmed in a brief interaction with a typically developing peer which will be coded to obtain social interaction skills and fluency scores.

SECONDARY OUTCOMES:
Change from Baseline Strengths and Difficulties Questionnaire (SDQ) after Intervention | One Week Post-Intervention
  The SDQ is a 25 item survey that asks about positive and negative attributes.
Change from Baseline Loneliness Scale after Intervention | One Week Post Intervention
  The Loneliness Scale is a 24-item survey that assesses social and emotional loneliness.
Change from Baseline Multidimensional Anxiety Scale for Children after Intervention | One Week Post-Intervention
  The MASC is a 39-item survey that assesses anxiety symptoms in children.
Change from Baseline Strengths and Difficulties Questionnaire (parent form)after Intervention | One Week Post-Intervention
  The Strengths and Difficulties Questionnaire is a 25 item survey that asks about positive and negative attributes.
Change from Baseline Strengths and Difficulties Questionnaire at 3 month Follow Up | 3 Month Follow Up
Change from Baseline Loneliness Scale at 3-month Follow Up | 3 Month Follow Up
Change from Baseline Multidimensional Anxiety Scale for Children at 3 month Follow Up | 3 Month Follow Up
Change from Baseline Strengths and Difficulties Questionnaire (parent form)at 3 Month Follow Up | 3 Month Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Murray, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Psychiatry Clinic, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No